CLINICAL TRIAL: NCT00654199
Title: Ventricular Asynchrony in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0507007970
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Ventricular Asynchrony in Cardiac Surgery Patients
Keywords: CABG; Ventricular Asynchrony; Normal Sinus Rhythm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

1. assess the existence of inter-ventricular and intra-ventricular asynchrony in cardiac surgery patients before (PRE) and after cardiopulmonary bypass surgery (POST)
2. investigate whether a modification of usual pacing practices (RA-LV pacing) can achieve inter- and intra-ventricular synchrony and improve heart function, as evaluated by hemodynamic and echocardiographic indexes, when compared with the patient's native rhythm (normal sinus rhythm (SR), or conventional pacing modes

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac surgery, in normal sinus rhythm

Exclusion Criteria:

* atrial fibrillation, abnormal hearth rhythms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States